CLINICAL TRIAL: NCT05727878
Title: A Study to Evaluate Safety and Efficacy of KPI-012 Ophthalmic Solution in Participants With Persistent Corneal Epithelial Defect (PCED)
Brief Title: Trial to Evaluate Safety and Efficacy of KPI-012 Ophthalmic Solution in Participants With PCED
Acronym: CHASE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Combangio, Inc (Industry)
Collaborators: Kala Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kala Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPI-012-C-001
Record Dates: First submitted 2023-02-06; First posted 2023-02-14 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Persistent Corneal Epithelial Defect

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Cohort 1: open-label Cohort 2: masked to participant, Investigator, site staff, outcomes assessor, etc
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1, Arm 1 (Experimental): KPI-012 High Dose KPI-012 Ophthalmic Solution 3 U/mL 1 drop 4 times/day for 56 days
  Interventions: Drug: KPI-012
- Cohort 2, Arm 1 (Experimental): KPI-012 Low Dose KPI-012 Ophthalmic Solution 1 U/mL 1 drop 4 times/day for 56 days
  Interventions: Drug: KPI-012
- Cohort 2, Arm 2 (Experimental): KPI-012 High Dose KPI-012 Ophthalmic Solution 3 U/mL 1 drop 4 times/day for 56 days
  Interventions: Drug: KPI-012
- Cohort 2, Arm 3 (Placebo Comparator): KPI-012 Vehicle KPI-012 Ophthalmic Solution 0 U/mL 1 drop 4 times/day for 56 days
  Interventions: Drug: KPI-012 Vehicle

INTERVENTIONS:
Drug: KPI-012 — KPI-012 is a secretome product composed of biologically active components secreted from human bone marrow-derived mesenchymal stem cells
  Arms: Cohort 1, Arm 1; Cohort 2, Arm 1; Cohort 2, Arm 2
Drug: KPI-012 Vehicle — KPI-012 formulation with no active drug
  Arms: Cohort 2, Arm 3

SUMMARY:
The primary objective of the study is to investigate the safety and efficacy of KPI-012 compared to vehicle in participants who have a documented clinical diagnosis of PCED.

DETAILED DESCRIPTION:
Approximately 90 participants diagnosed with persistent corneal epithelial defect (PCED) will be enrolled at multiple US centers in a study to assess the safety and efficacy of KPI-012, a topical mesenchymal stem cell secretome therapy. After an initial cohort of at least 2 participants to evaluate the safety of the high strength product, participants in the second cohort will be randomized to treatment with either the product or vehicle (placebo) for 8 weeks. The percentage of healing will be compared between groups treated with product and vehicle. Total length of study participation will be approximately 34 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Have PCED for at least 7 days prior due to an underlying condition such as diabetic keratopathy, herpetic eye disease, severe dry eye disease, limbal stem cell deficiency, infectious keratitis, neurotrophic keratitis, post ocular surgery, medical trauma, chemical burn, etc.
2. PCED measurements meet study criteria.

Exclusion Criteria:

1. Any active ocular infection or any active infectious disease that could impact the PCED.
2. Severe corneal burns in the Study Eye.
3. Severe limbal stem cell deficiency in either eye.
4. The circumference affected by limbal blood vessel ischemia greater than 75% of the circumference in the Study Eye.
5. Severe blepharitis or severe meibomian gland disease.
6. Severe eyelid abnormalities in the Study Eye, contributory to the persistence of the PCED.
7. Evidence of corneal ulceration.
8. Anticipated need for punctal occlusion.
9. Use of Oxervate in the Study Eye within past 30 days.
10. History of any surgical procedure for treatment of the study PCED.
11. History of any other ocular surgery in the Study Eye within 90 days prior to screening.
12. Not willing to suspend use of contact lens in the Study Eye.
13. Any use of Botox injections to induce pharmacologic blepharoptosis in the 90 days.
14. Expected use of systemic doxycycline.
15. Any use of chemotherapeutic agents within 7 days prior to Study, or anticipated use during the study.
16. History of current drug or alcohol abuse or addiction.
17. Use of another investigational agent within 30 days.
18. Participants who are pregnant, breastfeeding, or planning a pregnancy during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-10-19 (Actual)

PRIMARY OUTCOMES:
Response status | Day 56
  Complete healing of the PCED and no corneal fluorescein staining in the area of the study lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Veasey, Study Director — Kala Pharmaceuticals, Inc.
Locations (41):
- United States (38):
  - Principal Investigator, Dothan, Alabama
  - Principal Investigator, Irvine, California
  - Principal Investigator, La Jolla, California
  - Principal Investigator, Loma Linda, California
  - Principal Investigator, Los Angeles, California
  - Principal Investigator, Pasadena, California
  - Principal Investigator, Rancho Cordova, California
  - Principal Investigator, Aurora, Colorado
  - Principal Investigator, Fort Collins, Colorado
  - Principal Investigator, Littleton, Colorado
  - Principal Investigator, Miami, Florida
  - Principal Investigator, Orange City, Florida
  - Principal Investigator, Atlanta, Georgia
  - Principal Investigator, Carmel, Indiana
  - Principal Investigator, Indianapolis, Indiana
  - Principal Investigator, Louisville, Kentucky
  - Principal Investigator, Boston, Massachusetts
  - Principal Investigator, Chesterfield, Missouri
  - Principal Investigator, Kansas City, Missouri
  - Principal Investigator, St Louis, Missouri
  - Principal Investigator, Palisades Park, New Jersey
  - Principal Investigator, New York, New York
  - Principal Investigator, Rockville Centre, New York
  - Principal investigator, Durham, North Carolina
  - Principal Investigator, Garner, North Carolina
  - Principal Investigator, Powell, Ohio
  - Principal Investigator, Philadelphia, Pennsylvania
  - Principal Investigator, Pittsburgh, Pennsylvania
  - Principal Investigator, Rapid City, South Dakota
  - Principal Investigator, Memphis, Tennessee
  - Principal Investigator, Nashville, Tennessee
  - Principal Investigator, Austin, Texas
  - Principal Investigator, Houston, Texas
  - Principal Investigator, San Antonio, Texas
  - Principal Investigator, Norfolk, Virginia
  - Principal Investigator, Seattle, Washington
  - Principal Investigator, Morgantown, West Virginia
  - Principal Investigator, Kenosha, Wisconsin
- Argentina (2):
  - Principal Investigator, Caba, Buenos Aires
  - Principal Investigator, Rosario, Santa Fe Province
- Principal Investigator, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No